CLINICAL TRIAL: NCT06395506
Title: An Open-label Randomized Trial of Exercise ± Creatine Supplementation to Augment the Adaptations of Exercise Training in Cancer Survivors
Brief Title: THRIVE Well Cancer FDTN/Exercise_Creatine Supplementation
Acronym: THRIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: ThriveWell Cancer Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-0215
Record Dates: First submitted 2024-04-19; First posted 2024-05-02 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Breast Cancer Female; Muscle Weakness
Keywords: Breast Cancer; Breast Cancer Female; Exercise; Creatine Supplement
MeSH Terms: conditions — Breast Neoplasms; Muscle Weakness; Motor Activity | interventions — Creatine

STUDY DESIGN:
Intervention Model Description: This study plans to enroll 30 breast cancer patients who have completed chemotherapy within 6 months prior to consenting for this study. Each arm will have 15 participants. One arm will receive creatine and the other will serve as the control group with no creatine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Age-Matched Control Group (No Intervention): Women who have never been diagnosed with cancer.
- Creatine Supplement Group (Experimental): Those randomized to receive creatine (experimental group) will be initially dosed at 20 g/day for 7 days to boost availability of creatine systemically. Thereafter, the dose will be reduced to 5 g/day for maintenance through the duration of the 12-week protocol. Participants will engage in three center-based exercise sessions each week for 12 weeks; each session lasting roughly 1-hour. Participants will be given a fitbit (electronic watch that measures steps or heart rate) as well to track heart rate and monitor activity throughout the study.
  Interventions: Dietary Supplement: Creatine
- Non-Creatine Supplement Group (No Intervention): Participants will engage in three center-based exercise sessions each week for 12 weeks; each session lasting roughly 1-hour. Participants will be given a Fitbit (electronic watch that measures steps or heart rate) as well to track heart rate and monitor activity throughout the study.

INTERVENTIONS:
Dietary Supplement: Creatine — Those randomized to receive creatine (experimental group) will be initially dosed at 20 g/day for 7 days to boost availability of creatine systemically. Thereafter, the dose will be reduced to 5 g/day for maintenance through the duration of the 12-week protocol.
  Arms: Creatine Supplement Group

SUMMARY:
The study's purpose is to evaluate whether creatine supplementation can help breast cancer survivors respond quicker to exercise by improving strength, endurance, and body composition. We are seeking to compare information collected from healthy woman of the same age who have never had breast cancer to those participants who have had breast cancer and undergone chemotherapy treatment.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the effects of creatine supplementation in modulating strength and physical function in breast cancer survivors that have recently completed chemotherapy. The primary objective is to determine the effects of creatine in modulating strength and physical function in cancer survivors.

ELIGIBILITY:
Inclusion criteria (Breast Cancer Group)

* Age 18-75 years of age
* Diagnosis of breast cancer requiring chemotherapy
* Recent (within 6 months) completion of chemotherapy
* Willing to attend 3 virtual-based exercise sessions per week
* Able to take oral medications
* Participant is willing and able to provide consent to participating in the study
* Serum creatinine ≤ 1.5 x ULN or Estimated glomerular filtration rate (eGFR) ≥30 mL/min/1.73 m2 by Chronic Kidney Disease Epidemiology Collaboration equation.

Exclusion criteria (Breast Cancer Group)

* Physical indications where performing exercise may be limited and/or contraindicated
* Poorly controlled hypertension (blood pressure > 160/95mmHg)
* Current tobacco use (within 6 months)
* Anabolic steroids use
* Pitting edema greater than 2+
* Currently undergoing chemotherapy treatment for cancer
* History of moderate-severe heart disease (New York Heart Classification greater than grade II) or pulmonary disease (dyspnea on exertion upon climbing one flight of stairs or less; abnormal breath sounds on auscultation)
* Pregnant or plan to become pregnant during the study
* Recent (within one month) or anticipated treatment with corticosteroids (except for short term use during the time of chemotherapy), or other appetite stimulants
* Serum creatinine > 1.5 x ULN or Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 by Chronic Kidney Disease Epidemiology Collaboration equation
* Currently taking creatine supplements
* Lack of availability to a smartphone and/or internet

Inclusion Criteria (Healthy Age-matched Control Group)

* Age 18-75 years of age
* Have never been diagnosed with cancer
* Willing to provide consent to participate in this study

Exclusion Criteria (Healthy Age-matched Control Group)

* Physical indications where performing exercise may be limited and/or contraindicated
* Poorly controlled hypertension (blood pressure > 160/95mmHg)
* Current tobacco use (within 6 months)
* Anabolic steroids use
* Pitting edema greater than 2+
* History of cancer diagnosis
* History of moderate-severe heart disease (New York Heart Classification greater than grade II) or pulmonary disease (dyspnea on exertion upon climbing one flight of stairs or less; abnormal breath sounds on auscultation)
* Pregnant or currently taking prescribed medication to prepare for pregnancy (i.e.

hormonal therapy for IVF)

* Recent (within one month) treatment with corticosteroids
* Recent (within one month) use of appetite stimulants or appetite suppressants
* Serum creatinine > 1.5 x ULN or Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 by Chronic Kidney Disease Epidemiology Collaboration equation
* Diagnosed Bipolar Disorder or MDQ score indicative of bipolar disorder or Neurological disorders
* Uncontrolled diabetes (A1c of 6.5% or higher)
* Currently taking creatine supplements
* Lack of availability to a smartphone and/or internet

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in strength in breast cancer survivors | baseline and 12 weeks
  Determine the change in strength in breast cancer survivors by comparing pre and post measurements of strength measurement tools including 1RM/10RM/Biodex evaluations.
Change in physical functional capacity in breast cancer survivors | baseline and 12 weeks
  Determine the change in strength in breast cancer survivors by comparing pre and post measurements of the six minute walk test.

SECONDARY OUTCOMES:
Change intramuscular storage of creatine | baseline and 12 weeks
  Determine the change in intramuscular storage of creatine by comparing pre and post vastus lateralis muscle using MRI.
Change in body composition in cancer survivors | baseline and 12 weeks
  Determine the change in body composition in breast cancer survivors by pre and post measurements of bone mass as well as lean vs fat mass via a DEXA scan.
Change in the return of strength for breast cancer survivors with creatine + exercise | 12 weeks
  Breast cancer survivors who complete 12-weeks of exercise with creatine supplementation group who regained strength and physical function to that of women of similar age who never had cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Darpan Patel, PhD, Principal Investigator — University of Texas
Locations (1):
- The University of Texas Medical Branch, Galveston, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No